CLINICAL TRIAL: NCT00387270
Title: A Multicenter, Phase 1-2A, Open-Label, Dosage-Escalation and Randomized, Double-Blinded, Placebo-Controlled Study of Dimebon in Subjects With Huntington's Disease
Brief Title: Safety Study of the Novel Drug Dimebon to Treat Patients With Huntington's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medivation, Inc. (Industry)
Collaborators: Huntington Study Group (Network)
Responsible Party: Karl Kieburtz, MD, Clinical Trial Coordination Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIM03; DIMOND
Record Dates: First submitted 2006-10-10; First posted 2006-10-12 (Estimated); Last update posted 2008-01-04 (Estimated); Status verified 2007-09

CONDITIONS: Huntington's Disease
Keywords: Huntington's disease; Dimebon; dose-escalation; Phase 1-2a; randomized; controlled; double-blind; Unified Huntington's Disease Rating Scale
MeSH Terms: conditions — Huntington Disease | interventions — latrepirdine

ARMS (1):
- A (Experimental): Dimebon
  Interventions: Drug: Dimebon

INTERVENTIONS:
Drug: Dimebon — Dimebon 10 or 20 mg TID x 7 days

SUMMARY:
This study is being conducted to determine the safety and tolerability of Dimebon in people with Huntington's disease after short-term exposure (one week) and after longer exposure (three months). Also, the study will assess whether or not there is an effect of Dimebon on the symptoms of Huntington's disease, including cognitive (thinking abilities), motor (movement), behavior, and overall functioning.

ELIGIBILITY:
Inclusion Criteria:

* Clinical features of Huntington's disease and a confirmatory family history of HD, or a CAG repeat expansion greater than or equal to 36
* Stage I,II,III HD and a total functional capacity greater than or equal to 5 on the Unified Huntington's Disease Rating Scale

Exclusion Criteria:

* Clinical evidence of unstable medical illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-10; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities | 7 days

SECONDARY OUTCOMES:
Unified Huntington's Disease Rating Scale | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Karl D Kieburtz, MD, Principal Investigator — University of Rochester Medical School, Huntington Study Group
Locations (1):
- Huntington Study Group, Rochester, New York, United States

REFERENCES:
- See also: The Huntington Study Group (HSG) is a non-profit group of physicians and other health care providers from medical centers in the U.S., Canada, Europe, and Australia, experienced in the care of Huntington patients and dedicated to clinical research of HD — http://www.huntington-study-group.org